CLINICAL TRIAL: NCT04412564
Title: A Open-label, Single-arm Phase Ⅱ Clinical Trial of TQ-B3101 Capsules in Subjects With Advanced Malignant Tumor
Brief Title: A Study of TQ-B3101 Capsules in Subjects With Advanced Malignant Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3101-II-03
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3101 capsules (Experimental): TQ-B3101 capsules 300mg bid administered orally in 28-day cycle.
  Interventions: Drug: TQ-B3101

INTERVENTIONS:
Drug: TQ-B3101 — TQ-B3101 is a ALK inhibitor.

SUMMARY:
The objective of this study is to evaluate efficacy and safety of TQ-B3101 in subjects with advanced malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

-1. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; Life expectancy ≥12 weeks.

2. Understood and signed an informed consent form. 3. Histologically or cytologically confirmed advanced malignant solid tumors. 4. Adequate organ system function. 5. Patients need to adopt effective methods of contraception.

Exclusion Criteria:

* 1. Has multiple factors affecting oral medication. 2. The toxicity of previous antitumor treatment is not recovered to ≤ grade 1. 3. Other malignancies occurred within 3 years, with exception of cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors.

  4. Has a history of hypertension, hypertensive encephalopathy or uncontrolled hypertension.

  5. Has cardiovascular and cerebrovascular diseases. 6. Has received radiotherapy, chemotherapy, surgery less than 4 weeks before the first dose.

  7. Has central nervous system metastasis and / or spinal cord compression, cancerous meningitis, and meningeal disease.

  8. Active hepatitis, HIV positive, syphilis positive. 9. Has a history of psychotropic substance abuse. 10. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Adverse events (AE) and serious adverse events (SAE) | up to 48 weeks
  The occurrence of all adverse events (AE) and serious adverse events (SAE).

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 48 weeks
  PFS defined as the time from first dose until the first documented progressive disease (PD) or death from any cause.
Disease control rate (DCR) | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Overall survival (OS) | up to 48 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (36):
- China (36):
  - Anhui Chest Hospital, Hefei, Anhui
  - The Second Hospital of Anhui medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA Ceneral Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - Luoyang Central Hospital Affiliated to Zhenghzou University, Luoyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang First People's Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Weihai Central Hospital, Weihai, Shandong
  - Shanghai Jiaotong University Affiliated Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethuen Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an Chest Hospital, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Kashgar Prefecture, Kashgar Prefecture, Xinjiang Uygur Autonomous Region
  - First Affiliated Hospital, School of Medicine, Shihezi University, Shihezi, Xinjiang Uygur Autonomous Region
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang